CLINICAL TRIAL: NCT02188654
Title: Metformin: A Valid Add-On Drug in the Treatment of Psoriatic Arthritis-Randomized Controlled Trial
Brief Title: Metformin in Psoriatic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, MD, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: alexmed12671416
Record Dates: First submitted 2014-07-04; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; inflammation; metabolic syndrome; metformin
MeSH Terms: conditions — Arthritis, Psoriatic; Inflammation; Metabolic Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): 500 mg metformin
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 500 mg of placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — 500mg/day retarded formulation of metformin
  Arms: Metformin
Drug: Placebo — 500 mg/day of placebo tablets
  Arms: Placebo

SUMMARY:
Psoriatic arthritis (PsA) is a systemic, inflammatory disease. The chronic inflammation in PsA predisposes patients to the metabolic syndrome (MetS). MetS is associated with systemic inflammation and proinflammatory cytokines. Clinical observations and experimental results argue for an anti-inflammatory and immunosuppressant property of MET.

DETAILED DESCRIPTION:
The chronic inflammatory nature of psoriasis and PsA predisposes patients to cardiovascular diseases and metabolic syndrome (MetS). MetS is associated with systemic inflammation and proinflammatory cytokines.Clinical observations and experimental results argue for an anti-inflammatory and immunosuppressant property of MET.

A randomized placebo-controlled trial was conducted to evaluate the efficacy and safety of metformin as add-on therapy to MTX compared to MTX after 24 weeks in patients with PsA.

The study randomized 56 patients with a diagnosis of PsA . Patients with a history of a cardiovascular event and diabetics were excluded. Body mass index (BMI) and classic cardiovascular risk factors were recorded. Blood samples were analysed for glucose, lipid profile, ESR, hsCRP, proinflammatory cytokines; tumour necrosis factor alpha (TNF-alpha), interleukin-6 (IL-6) and IL-17. The homeostasis model assessment model for insulin resistance (HOMA-IR) was used. The patients were randomized in a 1:1 ratio to receive 500mg/day retarded formulation of metformin (n=29) or placebo (n=29). Continuation of stable doses of MTX (25mg/week), NSAIDs, and/or corticosteroids (prednisone <10 mg/day) was permitted. Metformin drug pause on the day of MTX was given. Folic acid supplementation was given to both groups. The primary clinical endpoint was the ACR 20% (ACR20) response at 24 weeks. Secondary endpoints included reduction in PASI score, Health Assessment Questionnaire- Disability Index (HAQ-DI) and Psoriatic arthritis response criteria (PsARC) score.

ELIGIBILITY:
Inclusion Criteria:

* Psoriatic arthritis patients

Exclusion Criteria:

* other inflammatory conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
ACR20 response | 24 weeks

SECONDARY OUTCOMES:
PASI score | 24 weeks
Health Assessment Questionnaire | 24 weeks
Disability Index (HAQ-DI) | 24 weeks
Psoriatic arthritis response criteria (PsARC) score | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD, Principal Investigator — University of Alexandria
Locations (1):
- University of Alexandria, Alexandria, Alexandria Governorate, Egypt